CLINICAL TRIAL: NCT06550206
Title: The Malleability of Social Group Understanding in Infancy and Early Childhood
Brief Title: Toddlers' Responses to Strangers
Status: Recruiting | Type: Observational
Sponsor: University of California Santa Cruz (Other)
Collaborators: New York University (Other); University of Maryland, College Park (Other)
Responsible Party: Sponsor
Other Study IDs: HS-FY2023-23
Record Dates: First submitted 2024-08-06; First posted 2024-08-12 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Social Behavior
MeSH Terms: conditions — Social Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Children's stranger wariness response to strangers — Children will see two strangers, one from a familiar racial background and one from an unfamiliar racial background. Familiar race stranger will be from the same racial background as the child's caregiver and unfamiliar race stranger will not.
  Other Names: Social bias

SUMMARY:
The study will assess if toddlers show differences in stranger wariness according to race, temperament, social network diversity, and neighborhood diversity.

DETAILED DESCRIPTION:
This study is investigating 13- to 24-month-old toddlers' reactions to meeting new people from familiar and unfamiliar racial backgrounds! Participation involves a 1-hour one-time visit to the researcher's lab, located on the UC Santa Cruz campus.

The study itself will take about 20 minutes, but will ask for a 1-hour visit to make sure child participants feel comfortable in the new space. The study will video record as child participants interact with two adults, who will play with the child and offer toys. Parent participants will also be asked to complete two surveys, one demographic survey and one social network survey, so that investigators can better understand how the people children see in their daily lives relate to how participants react to strangers from different racial backgrounds.

ELIGIBILITY:
Inclusion Criteria:

* typically developing
* age 13-24 months

Exclusion Criteria:

- any known developmental delays

Ages: 13 Months to 24 Months | Sex: All
Age Groups: Child
Study Population: Community sample from the larger Santa Cruz area
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Social Wariness | Through study completion, an average of 10 years
  children's social wariness as assessed by the time that the child first vocalized, touched the stranger, and the duration of time that the child stayed near their parent in seconds standardized and averaged to create a composite score.
Social Preference | Through study completion, an average of 10 years
  Social preference will be coded by observing toddler behavior and assigning the following codes: 1 = did not take the toy from either stranger, 2 = took toy from familiar race stranger, 3 = took toy from unfamiliar race stranger, 4 = took toy or played with both strangers simultaneously.

CONTACTS AND LOCATIONS:
Overall Officials: Hyesung Hwang, PhD, Principal Investigator — University of California Santa Cruz
Locations (1):
- Social Science 2 Building, Santa Cruz, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All anonymized IPD data that underlie a publication will be shared after the study is published on open science framework.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available within a period of 10 years. Anonymized aggregate data will be available indefinitely. No identifiable data will be shared.
Access Criteria: All anonymized data will be available once study has been published and will be available indefinitely.

REFERENCES:
- [Background] Hwang HG, Filippi CA, Morales S, Fox NA, Woodward A. Children's social wariness toward a different-race stranger relates to individual differences in temperament. Dev Sci. 2023 Nov;26(6):e13390. doi: 10.1111/desc.13390. Epub 2023 Mar 24. PMID 36960937